CLINICAL TRIAL: NCT01346007
Title: Study of Safety, Immunogenicity and Immunological Memory of 7-valent Pneumococcal Conjugate Vaccine in Children With Idiopathic Nephrotic Syndrome
Brief Title: Study of 7-valent Pneumococcal Conjugate Vaccine in Children With Idiopathic Nephrotic Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Dr Vana Spoulou, 1st Department of Pediatrics, Division of Infectious Diseases 'Aghia Sophia' Children's Hospital, Athens University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NKU 7049687
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2009-01

CONDITIONS: Idiopathic Nephrotic Syndrome
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Active Comparator): Children with idiopathic nephrotic syndrome in remission treated with low-dose prednisolone and/or mycophenolate mofetil and/or cyclosporine A
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine
- controls (Active Comparator)
  Interventions: Biological: 7-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugate vaccine — A 0,5 ml dose of 7-valent pneumococcal conjugate vaccine in both arms A 0,5 ml anamnestic dose of 7-valent pneumococcal conjugate vaccine in subjects with idiopathic nephrotic syndrome 12 months after priming
  Other Names: Prevenar; Wyeth Vaccines

SUMMARY:
The purpose of this study is to determine whether 7-valent pneumococcal conjugate vaccine safely induces immune responses and immunological memory in children with idiopathic nephrotic syndrome in remission.

DETAILED DESCRIPTION:
Idiopathic nephrotic syndrome (INS) is the most frequent glomerular disease in children under 16 years old with incidence rate 2-7/100,000 patients/year depending on ethnicity. Those patients are susceptible to invasive pneumococcal disease (IPD) including peritonitis, pneumonia with or without pleural effusion and meningitis. Due to increased mortality and risk of relapses associated with IPD, it has been recommended that children with INS should be immunized with pneumococcal conjugate vaccine [1]. However, concerns on vaccine safety and impaired immunogenicity due to INS pathogenesis and immunosuppressive treatment are a hurdle for universal implementation of existing guidelines.

To thoroughly evaluate safety of 7-valent pneumococcal conjugate vaccine (PCV7) in children with INS in remission, we will investigate a possible association of vaccination with increased risk for recurrences of INS. We will also study immunogenicity and kinetics of immune response in INS patients and healthy subjects and the effect of different types of treatment on primary immune response and antibody persistence at 12-14 months following vaccination with PCV7.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Between 2-20 years of age

Exclusion Criteria:

* serious allergic reaction to previous vaccination
* history of invasive pneumococcal disease
* vaccination with pneumococcal conjugate vaccine
* vaccination with pneumococcal polysaccharide vaccine
* administration of intravenous immunoglobulin or other blood products during the last 3 months

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Pneumococcal serotype-specific antibodies and B memory cells | Within the first 30 days after vaccination

SECONDARY OUTCOMES:
Incidence of relapses of idiopathic nephrotic syndrome | Within 12 months after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Maria Theodoridou, Dr, Study Chair — 1st Department of Pediatrics, Division of Infectious Diseases 'Aghia Sophia' Children's Hospital, Athens University School of Medicine; Vana Spoulou, Dr, Study Director — 1st Department of Pediatrics, Division of Infectious Diseases 'Aghia Sophia' Children's Hospital, Athens University School of Medicine; Christina Liakou, MD, Principal Investigator — 1st Department of Pediatrics, Division of Infectious Diseases 'Aghia Sophia' Children's Hospital, Athens University School of Medicine
Locations (1):
- 1st Department of Pediatrics, Division of Infectious Diseases 'Aghia Sophia' Children's Hospital, Athens University School of Medicine, Goudi, Athens, Greece